CLINICAL TRIAL: NCT04390516
Title: Prediction Of Respiratory Decompensation In Covid-19 Patients Using Machine Learning: The READY Trial
Brief Title: Respiratory Decompensation and Model for the Triage of COVID-19 Patients
Acronym: READY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dascena (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 051420
Record Dates: First submitted 2020-05-14; First posted 2020-05-15 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: COVID-19; Coronavirus; Mortality; Mechanical Ventilation
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COViage (Other): Machine learning intervention
  Interventions: Device: COViage

INTERVENTIONS:
Device: COViage — The COViage machine learning algorithm is designed to predict mechanical ventilation and mortality within 24 hours after hospital admission.

SUMMARY:
The purpose of this study is to prospectively evaluate a machine learning algorithm for the prediction of outcomes in COVID-19 patients.

DETAILED DESCRIPTION:
In a multi-center prospective clinical trial, a machine learning algorithm was deployed at five partner hospitals to analyze live patient data, including blood pressure and Creatinine levels, to determine the algorithm's ability to predict COVID-19 patient prognosis. The primary endpoint was mechanical ventilation of study subjects within 24 hours after hospital admission separate from a decompensation alert related to oxygen levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Confirmed COVID-19 infection through RT-PCR test

Exclusion Criteria:

* Patients aged less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Mechanically ventilated patient outcome | Through study completion, an average of 2 months
  Ventilated or not ventilated within 24 hours

SECONDARY OUTCOMES:
Mortality or mechanically ventilated patient outcome | Through study completion, an average of 2 months
  Death or ventilated, or no death or not ventilated within 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Dascena, Oakland, California, United States